CLINICAL TRIAL: NCT04061811
Title: Soluble Neprilysin, NT-proBNP, and Growth-Differentiation-Factor-15 as Biomarkers for Heart Failure in Dialysis Patients
Acronym: SONGBIRD
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); F-CRIN (Unknown)
Responsible Party: Principal Investigator, Michael Sören Balzer, Postdoctoral fellow, Hannover Medical School
Other Study IDs: 7952_BO_S_2018; KlinStrucMed program (Other Grant/Funding Number: Else Kröner-Fresenius-Stiftung)
Record Dates: First submitted 2019-08-16; First posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Heart Failure; End Stage Renal Disease
Keywords: congestive heart failure (HF); biomarker; chronic kidney disease (CKD); hemodialysis (HD); peritoneal dialysis (PD); neprilysin (NEP); growth differentiation factor-15 (GDF15)
MeSH Terms: conditions — Heart Failure; Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma, serum, peritoneal dialysate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HF (heart failure): Patients with end stage renal disease requiring dialysis with reduced or preserved ejection fraction.
  Interventions: Diagnostic Test: Diagnostic biomarker study
- Control: Patients with end stage renal disease requiring dialysis without HF.
  Interventions: Diagnostic Test: Diagnostic biomarker study

INTERVENTIONS:
Diagnostic Test: Diagnostic biomarker study — Comparing circulating concentrations of NT-proBNP, GDF15, and neprilysin (NEP) along with NEP activity in patients with and without HF, as diagnosed by clinical parameters and post-dialysis echocardiography.

SUMMARY:
Objectives: The aim of this study is to determine whether growth differentiation factor-15 (GDF15) and circulating neprilysin (cNEP) improve the diagnosis of congestive heart failure (HF) in patients on dialysis.

Background: Dialysis patients are at increased risk of HF. However, diagnostic utility of NT-proBNP as a biomarker is decreased in patients on dialysis. GDF15 and cNEP are biomarkers of distinct mechanisms that may contribute to HF pathophysiology in such cohorts.

Methods: We compare circulating concentrations of NT-proBNP, GDF15, and cNEP along with NEP activity in patients on chronic dialysis without and with HF, as diagnosed by clinical parameters and post-dialysis echocardiography. We use correlation, linear and logistic regression as well as receiver operating characteristic (ROC) analyses.

ELIGIBILITY:
Inclusion Criteria:

* ESRD on either chronic hemodialysis (HD) or peritoneal dialysis (PD) for ≥3 months

Exclusion Criteria:

* previous switch of the type of renal replacement therapy from HD to PD or vice versa
* age <18 years
* pregnancy
* plasma exchange or apheresis in the past 6 months
* unipolar pacemaker
* history of whole extremity amputation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: End stage renal disease (ESRD) patients on chronic dialysis.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
HF diagnosis | Baseline (at study entry (diagnostic biomarker study))
  Diagnosis of HF

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Balzer, MD, Principal Investigator — Hannover Medical School
Locations (2):
- Inserm Umr S-942, Paris, France
- Hannover Medical School, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No